CLINICAL TRIAL: NCT01803828
Title: Phase IV Study on New Insights in Remodeling of Diabetic Cardiomyopathy: Gender Difference in Intramyocardial, Molecular and Neuroendocrine Assessment in Response to Chronic Inhibition of Cyclic GMP Phosphodiesterase 5A
Brief Title: REmodelling in Diabetic CardiOmapathy: Gender Response to PDE5i InhibiTOrs
Acronym: RECOGITO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Andrea M. Isidori, Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RECOGITO
Record Dates: First submitted 2013-02-26; First posted 2013-03-04 (Estimated); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Diabetic Cardiomyopathy; Diabetes Mellitus Type 2
Keywords: Diabetic Cardiomyopathy; Genders; Phosphodiesterase 5A inhibitors; endothelial dysfunction; inflammation; diabetic complications
MeSH Terms: conditions — Diabetic Cardiomyopathies; Diabetes Mellitus, Type 2; Inflammation; Diabetes Complications | interventions — Tadalafil

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- Drug Group (Tadalafil) (Active Comparator): Tadalafil 20 mg
  Interventions: Drug: Tadalafil
- Placebo Group (PLC) (Placebo Comparator): Placebo 20 mg
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tadalafil — 20 mg/die (1 capsule)
  Other Names: Cialis 20 mg
  Arms: Drug Group (Tadalafil)
Drug: Placebo — Placebo 20 mg/die (1 capsule)
  Arms: Placebo Group (PLC)

SUMMARY:
Pathophysiology of diabetic cardiomyopathy (DCM) is yet unclear and gender differences at baseline and a specific treatment have not been indicated. The investigators already demonstrated the positive impact of phosphodiesterase type 5A (PDE5A) inhibition in men. The investigators' study aims to characterize DCM, measuring molecular and neuroendocrine assessment to relate to intramyocardial metabolism and cardiac kinetic. The investigators will perform a randomized, placebo-controlled, double-blind study enrolling 164 diabetic patients (females and males) with DCM, to evaluate gender responses to 6 months of PDE5A inhibitors (PDE5Ai). The investigators' study will describe gender differences in DCM features. The proposed research will test whether PDE5Ai could become a new target for antiremodeling drugs and to discover a molecular pathways affected by this class of drugs and a network of circulating markers for the early diagnosis, monitoring and prediction of response to treatment of DCM.

DETAILED DESCRIPTION:
DCM is yet unclear and gender differences at baseline and a specific treatment have not been indicated. The study aims to characterize DCM, measuring molecular and neuroendocrine assessment to relate cardiac kinetic. The investigators will perform a randomized, placebo-controlled, double-blind study enrolling 120 diabetic patients with DCM, to evaluate gender responses to 5 months of PDE5Ai. The study will describe gender differences in DCM features. The proposed research will test whether PDE5Ai could become a new target for antiremodeling drugs and to discover a molecular pathways affected by this class of drugs and a network of circulating markers for the early diagnosis, monitoring and treatment of DCM.

In vitro studies have shown that phosphodiesterase 5 overexpression reduces cGMP levels and exacerbates remodeling. The investigators already studied the effects of 3-months daily Inhibition of cGMP hydrolysis through a phosphodiesterase 5A inhibitor (PDE5i) on cardiac remodeling in a cohort of asymptomatic, middle-aged men with type 2 diabetes mellitus (T2DM). CMR imaging revealed that diabetic cardiomyopathy in these patients produced an uncoupling in left ventricular contraction between longitudinal strain, which is reduced, and cardiac axial rotation, which is increased. Characterized DCM at early asymptomatic stages in men, we identified two circulating markers, TGF-beta and MCP-1 increased and significantly related to cardiac kinetic parameters. Then, the investigators found that long-term PDE5i restored coupling by reducing torsion and improving strain. It also reduced the ratio of left ventricular mass to end-diastolic volume that is increased in the presence of concentric hypertrophy. Circulating markers TGF-beta and MCP-1, significantly decreased after PDE5i vs. Placebo.These data suggest that phosphodiesterase 5 inhibition could work as an antiremodeling drug by acting directly on cardiac tissue, independently of other secondary vascular, endothelial, or metabolic effects.

However, these data need to be validated on a wide sample, for a longer duration of treatment, and including women, because of their high vulnerability to diabetic damage with preferential evolution in chronic heart failure, compared to males that frequently have ischemic complications.

T2DM is also considered a state of persistent inflammation that likely plays a role in development cardiovascular disease. Some studies have suggested that inflammation may impair the tissue repair process in diabetes, which appears delayed, unsupervised, and associated with higher levels of circulating classical monocytes.

The interaction between angiogenic cells and the endothelium is still critical for inflammatory cells to move and home in specific tissue sites in various pathological conditions. The Tie2 receptor is highly enriched in the endothelium and actively signals vascular quiescence. It is also expressed by in a unique subset of monocytes, Tie2-expressing monocytes (TEMs), which have been considered crucial for tissue remodeling and repair. Tie2 is stimulated by angiopoietin-1 (Ang1), a protein secreted by peri-endothelial cells and platelets. In the context of inflammation, a paralog of Ang1 called Ang2 competitively inhibits Tie2, normal endothelialcell function depends in part on a tightly regulated balance between Ang1 and Ang2. There is evidence of angiopoietin deregulation T2DM.

Several studies demonstrate that PDE5 inhibitors, have cardioprotective effects in different conditions, particularly in in diabetes. PDE5is reduce circulating inflammatory cytokines, protect against tissue damage, exert an anti-inflammatory response, preserve endothelial cell function and increase angiogenic mediators, including Ang1 in mouse models. The PDE5is also improves metabolism and these effects are extended to adipose tissue function.

Another diabetic complication is Diabetic polyneuropathy (DPN). DPN is characterized by loss and degeneration of neurons, Schwann cells, and neuronal fibers resulting in slowing of nerve conduction velocities.

cGMP is involved in the regulation of many neural functions, including neurotransmission, long term potentiation, gene expression, and even neurotoxicity and neurodegeneration. Hyperglycemia up-regulates PDE-5 in Schwann cells and reduces their proliferation and migration. Schwann cells play an important role in regenerating the peripheral nervous system by their capacity to proliferate, migrate, and secrete numerous factors that control nerve regeneration. Decreased proliferation of Schwann cells has also been demonstrated in both human and experimental models of diabetes. Therefore, reduction of cGMP levels by hyperglycemia suppresses Schwann cell proliferation and migration. Elevation of cGMP by blockage of PDE5 with sildenafil completely abolished and reverses the effect of hyperglycemia on Schwann cells in mice.

These changes are accompanied by change in serum neurotropic factors that are witnesses of active remodeling and regeneration at the neuronal level. Many studies in diabetic mice demonstrated that cGMP induces Schwann cells to synthesize nerve growth factor (NGF), neurotropic 3 (NT3) and BDNF.

One third of diabetes patients suffers from diabetic nephropathy (DN), a leading cause of end-stage renal disease. To date, effective treatment in halting or reversing the natural progression of DN remains uncertain. The pathophysiology is multifactorial and the molecular pathways involved are complex. Glomerular endothelial cell injury plays a major role in the development and progression of diabetic kidney disease, that is considered the result of converging hemodynamic and metabolic insults.

In kidney PDE5 is expressed in the glomeruli, mesangial cells, cortical tubules, inner medullary collecting duct and plays a critical role in the regulation of excretory function. In diabetes, glomerular cGMP production is decreased, PDE5 activity is increased and changes in the cGMP-NO pathway leads to a rise in intra-glomerular pressure.

PDE5 inhibitors may have an active role in the management of DN by reducing glomerulosclerosis and proteinuria and improving vascular inflammation and podocyte count in experimental diabetes models. These findings, together with the modulation of inflammatory and angiogenic mediators, and endothelial function in murine and human models, support the use of PDE5i to prevent complications of the diabetic kidney. Intriguingly, sildenafil, a potent PDE5i, was also associated with improved kidney function in patients with pulmonary arterial hypertension and in type-2 diabetes (T2DM) patients.

We hypothesize that:

* there are gender differences in left ventricular myocardial remodeling of T2DM patients detectable with tagged-CMR in terms of myocardial strain and ventricular torsion;
* gender-related features determine different cardiac response to PDE5i treatment detected by changes in ventricular contractility (strain and torsion on tagged-CMR);
* neuroendocrine (e.g. natriuretic peptides), metabolic markers, chemokines , circulating and cellular angiogenesis mediators might identify those asymptomatic patients at greatest risk of developing the diabetic complications (cardiomyopathy, neuropathy, nephropathy);
* neuroendocrine (e.g. natriuretic peptides), metabolic markers, chemokines , circulating and cellular angiogenesis mediators able to predict response to treatment with PDE5i and the evolution of diabetic complications;
* chronic treatment with PDE5i could restore or shut down neurological diabetic damage;
* chronic treatment with PDE5i could restore or shut down renal diabetic damage.

The aims of the study are:

Characterization of gender differences in DCM remodeling through a cluster of biomarkers indicative of the stage of the disease and CMR quantification of kinetic parameters (myocardial strain, ventricular torsion), fibrosis amount (T1-mapping technique).

Quantification of a cluster of biomarkers predictive of disease progression: metabolic and neuroendocrine markers, pro-fibrotic and pro-inflammatory circulating chemokines.

Evaluation of gender differences in the anti-remodeling effect of PDE5A inhibition in T2DM patients The investigators will perform a randomized, placebo-controlled, double-blind study enrolling 120 patients (females and males) with T2DM and diabetic cardiomyopathy. Patients will be randomized to treatment with PDE5Ai 20 mg / day or placebo for 5 consecutive months.

The outcomes will be evaluated before and 1 and 5 months after therapy.

Cardiovascular, endothelial and metabolic indices, and oxidative stress markers will be evaluated in all patients and related to CMR cardiac kinetic and metabolic parameters and fibrosis in order to identify:

* gender differences in kinetic parameters of left ventricle (end-diastolic volume, end-systolic volume, stroke volume, wall motion score index, myocardial strain, torsion angle, recoil rate with contraction dynamics);
* changes in myocardial fibrosis replacement amount (global contrast-enhanced T1 relaxation time, percentage of myocardial surface area, quantified by T1-mapping technique);

Diagnostic procedures will include:

* physical examination with measurement of anthropometric parameters (weight, waist circumference, hip circumference) and vital signs (blood pressure, heart rate);
* blood sampling for assessing glucose and lipid metabolism, liver, renal, hematopoietic and coagulative function, thyroid and androgen hormones, inflammatory parameters (cytokines, monocyte subpopulations);
* quantification of peripheral blood mononuclear cells (PBMC) subpopulations by flow cytometry;
* Circulating and cellular angiogenesis mediators assessment (angiogenic factors; cytokines, receptors and other angiogenic factors) by qRT-PCR and ELISA;
* SF36, FSFI (in women), IEFF e IPSS (in men) questionnaires, Infectious Diseases Questionnaire;
* cardiac exam, electrocardiogram and standard 2-D echocardiography with Tissue Doppler Imaging for diastolic function assessment and speckle tracking for cardiac kinetics measurement;
* assessment of body composition by a whole-body DEXA scan;
* magnetic resonance imaging (MRI) with contrast-enhanced cardiac tagging for evaluating kinetic parameters (torsion) and T1-mapping for assessing cardiac fibrosis;

Neurological examination to assess signs and symptoms related to polyneuropathy and autonomic neuropathy.

Specifically:

* evaluation of different sensitivity (diapason for vibratory, cotton wool for touch and pinprick for to pain);
* presence / reduction / absence of deep tendon reflexes;
* any motor deficits.

If any signs or symptoms consistent with diabetic neuropathy, to diagnosis confirm, these patients will undergo to a standard nerve conduction study for the large-caliber fibers (by registration of sensory potential stimulation from the sural, ulnar and radial nerve surface, and motors potential stimulation from peroneal and ulnar nerve). Those with large fiber neuropathy will be evaluate for small caliber fibers injuries with:

* evoked potentials laser;
* Quantitative Sensory Testing (QST);
* skin biopsy.
* renal doppler ultrasonography for the detection of possible renal complications through measurements of kidney volume and resistive index (RRI).

ELIGIBILITY:
Inclusion Criteria:

* age 45-80 years;
* Diagnosis of Type 2 Diabetes from at least 3 years;
* HbA1c < 10%;
* normal blood pressure or controlled hypertension;
* BMI < 40;
* SIV ≥ 11 mm men, ≥ 10 women and/or diastolic dysfunction (PW-doppler and TDI)

Exclusion Criteria:

* current use of PDE5 inhibitors;
* congenital or valvular cardiomyopathy;
* ischemic heart disease;
* proliferative retinopathy;
* contraindications to tadalafil use (hypersensitivity to tadalafil, nitrates use, severe cardiovascular disorders such as unstable angina or severe heart failure, severe hepatic impairment, blood pressure <90/50 mmHg, recent history of stroke or myocardial infarction and known hereditary degenerative retinal disorders such as retinitis pigmentosa);
* contraindications to CMR imaging with mdc (patients with implant such as cardiac pacemakers, insulin pumps, neurostimulators and cochlear implants, or metallic fragments, clips or devices, or severe renal failure with GFR < 30mL/min/1.73 m2);
* cronic or acute atrial fibrillation.

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Left Ventricular torsion (°) at 5 months | time 0, +5 months
  Change of Left ventricular torsion (°) assessed through CMR with tagging before and after treatment to heart failure and gender differences

SECONDARY OUTCOMES:
Change from baseline in cardiac shortening (Strain %) at 5 months | time 0, + 5 months
  Change of cardiac strain (%) and of parameters of cardiac geometry and performance assessed through CMR with tagging before and after treatment and gender differences
Change from baseline in Myocardial fibrosis at 5 months | time 0, +5 months
  Quantification of Myocardial fibrosis assessed with T1-mapping to establish a new parametersfor the characterization of DCM and treatment efficacy, assessed through CMR before and after treatment and gender differences
Change from baseline in Circulating pro-fibrotic and pro-inflammatory chemokines at 5 months | Time 0, +5 months
  Assessment of circulating pro-fibrotic and pro-inflammatory chemokines and correlation to torsion, strain and fibrosis at time 0 and after treatment (markers predictors of disease progression and treatment efficacy) and differences in genders
Peripheral immunological profile | time 0 and +5 months
  Evaluation of immune function and circulating and cellular angiogenesis mediators predictive of disease progression and PDE5Ai treatment efficacy
Gender differences in molecular, immunological and cardiac morpho-functional profile. | time 0 and +5 months
  Identify gender differences in molecular, immunological and imaging characterization of the DCM.
Effects of PDE5i on diabetic neuropathy | time 0 and +5 months
  Identify possible effects of chronic treatment with PDE5i on diabetic neuropathy
Effects of PDE5i on diabetic nephropathy | time 0 and +5 months
  Identify possible effects of chronic treatment with PDE5i on diabetic nephropathy
Effects of PDE5i on Body composition | time 0 and +5 months
  Evaluation of the effect of PDE5Ai on body composition evaluated by DEXA scan.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea M Isidori, MD, PhD, Principal Investigator — University of Roma La Sapienza
Locations (1):
- Dipartimento di Medicina Sperimentale - Sezione di Fisiopatologia Medica - Sapienza Università di Roma, Rome, Italy

REFERENCES:
- [Derived] Pofi R, Giannetta E, Feola T, Galea N, Barbagallo F, Campolo F, Badagliacca R, Barbano B, Ciolina F, Defeudis G, Filardi T, Sesti F, Minnetti M, Vizza CD, Pasqualetti P, Caboni P, Carbone I, Francone M, Catalano C, Pozzilli P, Lenzi A, Venneri MA, Gianfrilli D, Isidori AM. Sex-specific effects of daily tadalafil on diabetic heart kinetics in RECOGITO, a randomized, double-blind, placebo-controlled trial. Sci Transl Med. 2022 Jun 15;14(649):eabl8503. doi: 10.1126/scitranslmed.abl8503. Epub 2022 Jun 15. PMID 35704597